CLINICAL TRIAL: NCT04000581
Title: Does Increased Mobility Assessed With 3D Motion Tracking Technology Lead to Early Post-Operative Recovery Among Patients Undergoing Oncologic Surgeries
Brief Title: Impact of Early Mobility on Post-Surgery Recovery in Patients Undergoing Oncologic Surgeries
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty with equipment
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I 80918; NCI-2019-03139 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 80918 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2019-06-20; First posted 2019-06-27 (Actual); Results first posted 2021-08-31 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (usual care) (Active Comparator): Patients walk one to two laps around the ward twice per day, and have mobility tracked with Xsens over 5-10 minutes, until discharge from hospital. Patients also mobilize (walk out of the bed) on first day post-surgery under supervision and assistant of attending nurse in the floor if the clinical situation allows.
  Interventions: Other: Best Practice; Other: Questionnaire Administration
- Arm II (additional mobility) (Experimental): Patients walk for minimum 30 minutes per day and mobility is tracked with Xsens over 5-10 minutes up to discharge from hospital. Patients also mobilize (walk out of the bed) on first day post-surgery under supervision and assistant of attending nurse in the floor if the clinical situation allows.
  Interventions: Other: Physical Activity; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
  Arms: Arm I (usual care)
Other: Physical Activity — Walk for minimum 30 minutes per day
  Arms: Arm II (additional mobility)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies the impact of early mobility tracked with a 3-dimensional (3D) motion tracking technology (XSENS) on post-surgery recovery in patients undergoing oncologic surgeries. Xsens uses wireless measurements which could be used in clinical settings to objectively measure movement patterns (the joint range of movement and the distance of movement) during functional activities. Post-surgery mobility tracking may help doctors to identify the minimum required level of mobility after inpatient oncologic surgeries to enhance early post-surgery recovery and decrease early post-surgery complications.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate objectively using evidence based randomized controlled trial the impact of early mobility (first day after the surgery) after any inpatient oncologic procedures on early recovery of postoperative course.

II. Try to find out the minimum level of postoperative mobility that needed for early postoperative course recovery by objective assessment of range of movement for each participant using 3D motion tracking system (Xsens).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients walk one to two laps around the ward twice per day, and have mobility tracked with Xsens over 5-10 minutes, until discharge from hospital. Patients also mobilize (walk out of the bed) on first day post-surgery under supervision and assistant of attending nurse in the floor if the clinical situation allows.

ARM II: Patients walk for minimum 30 minutes per day and mobility is tracked with Xsens over 5-10 minutes up to discharge from hospital. Patients also mobilize (walk out of the bed) on first day post-surgery under supervision and assistant of attending nurse in the floor if the clinical situation allows.

After completion of study, patients are followed up for 30 days post discharge.

ELIGIBILITY:
Inclusion Criteria:

* Ambulant inpatient with a stay of >= 2 days after any inpatient oncologic surgery
* Eastern Cooperative Oncology Group (ECOG) scale of performance status of less than 3
* American Society of Anesthesiologist score (ASA) 3 or less
* Participants who do not engage in regular exercise regimen before the surgery (other than regular occupational physical therapy)
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Patients with altered mental status
* Patients with psychiatric illness
* ECOG scale performance status 3 or more
* ASA score of 4
* Participants who engage in regular exercise regimen before surgery (at least one session per week)
* Patients with restricted movement due to other diseases
* Patients who require continuous monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khurshid A Guru, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Usual Care) | Arm II (Additional Mobility)
Started | 5 | 12
Completed | 5 | 11
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Usual Care) | Arm II (Additional Mobility) | Total
Number analyzed (Participants) | 5 | 12 | 17
Age, Categorical [Count of Participants; unit: Participants] — Population: In the intervention arm, 2 patients have missing age. One patient removed their consent prior to any intervention.
  Participants
    number analyzed (Participants) | 5 | 10 | 15
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 3 | 4 | 7
    >=65 years | 2 | 6 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Two patients do not have age recorded.
  years
    number analyzed (Participants) | 5 | 10 | 15
    (all) | 63.2 (5.8) | 67.7 (8.4) | 66.2 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex was not recorded.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5 | 12 | 17
Godin Score [Mean (Standard Deviation); unit: units on a scale] — Godin Leisure Time Exercise Questionnaire Score
  * Designed to measure the level of sedentary behavior for an individual
  * The minimum score is 0 and the theoretical upper limit is 6,048
  * Higher values indicate more activity, while lower scores indicate sedentary activity. In general:
    1. <14 points = sedentary
    2. 14 - 23 points = moderately active
    3. 24 points or more = active Population: The baseline Godin Score was not obtained for 4 subjects.
  units on a scale
    number analyzed (Participants) | 4 | 9 | 13
    (all) | 21.3 (9.0) | 21.4 (12.0) | 21.3 (10.7)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Mobility
Description: changes in mobility (as measured by average velocity of pelvis) from baseline to discharge are compared between groups using a one-sided, two-sample t-test.
Time Frame: Baseline up to 30 days post discharge
Population: One patient (arm 2) removed consent prior to treatment initiation and outcome recording.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Arm I (Usual Care) | Arm II (Additional Mobility)
Number analyzed (Participants) | 5 | 11
m/s | 0.16 (0.15) | 0.58 (2.1)
Statistical Analysis 1: Comparison: Arm I (Usual Care) vs Arm II (Additional Mobility); The null hypothesis is that the mean change is equal between the groups, while the alternative is that an increased difference is observed in arm 2. The hypotheses are evaluated using a one-sided, two-sample t-test; Test type: Superiority; p = 0.329, t-test, 1 sided

2. Primary Outcome: Early Return of Bowel Motion
Description: Days from operation to passing flatus and/or stool, treated as continuous measure
Time Frame: Up to 30 days after discharge
Population: One patient (arm 2) removed consent prior to treatment initiation and outcome recording.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm I (Usual Care) | Arm II (Additional Mobility)
Number analyzed (Participants) | 5 | 11
days | 0.80 (0.45) | 0.90 (0.32)

3. Primary Outcome: Presence or Absence of Nausea and/or Vomiting
Description: Presence or absence of nausea and/or vomiting, treated as a binary variable
Time Frame: Up to 30 days after discharge
Population: Variable was not recorded.
Arm/Group | Arm I (Usual Care) | Arm II (Additional Mobility)
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Presence or Absence of Chest Symptoms
Description: Presence or absence of chest symptoms (cough, sputum, and ability of using incentive spirometry), treated as a binary variable
Time Frame: Up to 30 days after discharge
Population: Variable was not recorded.
Arm/Group | Arm I (Usual Care) | Arm II (Additional Mobility)
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Early Discharge From the Hospital
Description: Days from operation until hospital discharge, treated as continuous variable
Time Frame: Up to 30 days after discharge
Population: One patient (arm II) removed consent prior to treatment initiation and outcome recording.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm I (Usual Care) | Arm II (Additional Mobility)
Number analyzed (Participants) | 5 | 11
days | 2.0 (1.2) | 3.5 (2.8)

6. Primary Outcome: Surgical Related Complications and Readmissions
Description: Presence or absence of surgical complication (including readmission), treated as a binary variable
Time Frame: Up to 30 days after discharge
Population: Data were not collected.
Arm/Group | Arm I (Usual Care) | Arm II (Additional Mobility)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Range of Joint Movement in Upper and Lower Joints of Body
Description: Will be measured using the 3 dimensional (3D) motion tracking system (Xsens), to identify the minimum required level of mobility for better early postoperative course recovery.
Time Frame: Up to 30 days after discharge
Population: Data were not collected.
Arm/Group | Arm I (Usual Care) | Arm II (Additional Mobility)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Post-surgical Complications
Description: The complication status (present/absent) and grades will be summarized by group and compared using Fisher's exact test or the chi-square test, as appropriate.
Time Frame: Up to 30 days post discharge
Population: Data were not collected.
Arm/Group | Arm I (Usual Care) | Arm II (Additional Mobility)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in Exercise Habits Outside of the Hospital
Description: Post study questionnaire .
Time Frame: Up to 3 months post discharge
Population: This variable was not recorded.
Arm/Group | Arm I (Usual Care) | Arm II (Additional Mobility)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Application of Sensors in a Hospital Setting
Description: Adequate application of sensors, treated as a categorical variable
Time Frame: Up to 3 months post discharge
Population: One patient (arm 2) removed consent prior to treatment initiation and outcome recording.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Usual Care) | Arm II (Additional Mobility)
Number analyzed (Participants) | 5 | 11
Participants
  Adequate Sensor Application | 5 | 11
  Inadequate Sensor Application | 0 | 0

11. Secondary Outcome: Mobility Quality of Life Questionnaire
Description: The correlation between complication status and changes in mobility may be evaluated using a post study questionnaire.
Time Frame: Up to 3 months post discharge
Population: Data were not collected.
Arm/Group | Arm I (Usual Care) | Arm II (Additional Mobility)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Subjects will be followed 30 days post discharge to note any complications or readmission.
Arm/Group | Arm I (Usual Care) | Arm II (Additional Mobility)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/12
Other Adverse Events (participants affected / at risk) | 0/5 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT04000581/Prot_SAP_001.pdf
  • Informed Consent Form (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT04000581/ICF_000.pdf